CLINICAL TRIAL: NCT00756366
Title: Effects of Continuous Positive Airway Pressure Therapy on Myocardial Energetics and Sympathetic Nerve Function in Patients With Heart Failure and Obstructive Sleep Apnea.
Brief Title: CPAP Therapy in Patients With Heart Failure and Obstructive Sleep Apnea.
Acronym: PET-OSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Rob Beanlands, Robert S Beanlands, MD, FRCPC, Chief of Cardiology, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005982-01H; HSFO #NA5665; HSFO #T6426
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure; Obstructive Sleep Apnea
Keywords: positron emission tomography; myocardial energetics; sympathetic nerve function
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Heart Failure-OSA Group, randomized to early CPAP
  Interventions: Other: Positron Emission Tomography
- 2 (Active Comparator): Heart Failure-OSA Group, randomized to late CPAP
  Interventions: Other: Positron Emission Tomography
- 3 (Other): Heart Failure- no OSA, no CPAP therapy, observational group
  Interventions: Other: Positron Emission Tomography

INTERVENTIONS:
Other: Positron Emission Tomography — PET imaging at baseline, 1 week and 6-8 weeks. CPAP begins after baseline PET scan.
  Other Names: PET
  Arms: 1
Other: Positron Emission Tomography — PET imaging at Baseline, 1 week and 6-8 weeks. CPAP begins after 6-8 week PET scan.
  Other Names: PET
  Arms: 2
Other: Positron Emission Tomography — PET scan at baseline and 6-8 weeks, no CPAP therapy
  Other Names: PET
  Arms: 3

SUMMARY:
Heart failure affects approximately 5-6 million North Americans and is increasing in prevalence. Sleep-related disorders, such as obstructive sleep apnea (OSA) often coexist (11-37% incidence) with heart failure. OSA is the repeated temporary interruption of breathing during sleep and occurs when the air passages in the upper respiratory tract become blocked during sleep. OSA adversely affects the cardiovascular system resulting in hypoxia (decrease in oxygen supply), which decreases the oxygen supply to the heart. Patients with OSA are treated with continuous positive airway pressure (CPAP). It has also been shown that CPAP reduces angina during sleep, minimizes sympathetic nervous system (SNS) activation and improves left ventricular (LV) function, although the mechanism of action is not clear. Carbon-11 acetate PET imaging allows for the assessment of how the heart works and how efficiently the heart uses oxygen in certain circumstances. Carbon-11 hydroxyephedrine (HED) measures cardiac nervous system activity, which may have an effect on heart rate. The study will evaluate the term effects of continuous positive airway pressure (CPAP), a common treatment for patients with OSA, on the heart's efficiency or ability to work and its effect on the nervous system activity of the heart. Two patient groups will be evaluated 1.) patients with congestive heart failure and obstructive sleep apnea will be randomized to early or late CPAP to address the primary hypothesis of the study and 2.) patients with congestive heart failure only (matched control group). Both the primary randomized study group and secondary study group will be evaluated using [11C]acetate PET, [11C]HED PET and echocardiography. Measurements will be obtained at baseline, 1 week (where possible) and 6-8 weeks.

DETAILED DESCRIPTION:
OSA and heart failure (HF) are states of increased afterload, metabolic demand and sympathetic nervous system(SNS) activation. In patients with OSA and HF, CPAP initially may reduce LV stroke volume(SV) but subsequently improves LV function. This may relate to an early beneficial effect on myocardial energetics through early reduction in metabolic demand that subsequently leads to improved efficiency of LV contraction. However, it is not clear whether CPAP favourably affects cardiac energetics. Any such benefit may also relate to reduced SNS activation with CPAP therapy. However its effect on myocardial SN function is also not well studied. We propose to evaluate the temporal effect of CPAP on daytime 1) oxidative metabolism; 2) the WMI as an estimate of mechanical efficiency; 3) myocardial SN pre-synaptic function; and 4) HR variability in patients with OSA and HF. We will also determine whether these parameters are altered compared to a group of patients with HF without OSA. In conjunction with echocardiographic measures of LV stroke work, PET derived [11C]acetate kinetics will be used as a measure of oxidative metabolism, to determine the work metabolic index (WMI). [11C]HED retention will be used to measure cardiac SN pre-synaptic function.

HYPOTHESES

Primary Hypotheses:

In patients with chronic stable HF and OSA, 6-8 weeks' of CPAP demonstrates:

1. beneficial effects on daytime myocardial metabolism leading to a reduction in the rate of oxidative metabolism as measured by [11C]acetate kinetics using PET imaging;
2. improvement in energy transduction from oxidative metabolism to stroke work as measured by an increase in the daytime work-metabolic index.

Secondary Hypotheses:

In patients with chronic stable heart failure and OSA,

1. CPAP leads to an early (1 week'') reduction in daytime oxidative metabolism that precedes the improvement in work-metabolic index, indicating an early energy sparing effect;
2. CPAP leads to i) an increase in daytime myocardial SN pre-synaptic function as measured by increased [11C]HED retention on PET imaging, and ii) a parallel decrease in sympathetic and increase in vagal modulation of sino-atrial discharge (i.e. heart rate (HR) variability)
3. there is impaired daytime myocardial oxidative metabolism, work-metabolic index, and myocardial sympathetic nerve function compared to patients with heart failure without OSA.

'original protocol indicated 1 month follow up but was changed to 6-8 weeks in order to accommodate patient logistics and imaging centre scheduling.

''Logistics did not permit all patients to complete 1 week scan.

ELIGIBILITY:
Inclusion Criteria:

* systolic LV dysfunction (LVEF<40%; by echocardiography, radionuclide or contrast ventriculography)
* symptoms of HF: NYHA Class II to III
* stable condition with optimally tolerated medical therapy, unchanged for > 4 weeks
* Obstructive sleep apnea (OSA) diagnosed on nocturnal polysomnogram with an apnea/hypopnea index (AHI) >15 events/hr and a predominantly obstructive pattern(more than 80% of events being obstructive in nature)OR
* no OSA: defined as AHI<5 (control subjects) will be matched with the OSA group for gender, age + 5 years, ejection fraction (EF) +5%, drug therapy and etiology of HF (ischemic or non-ischemic)
* willingness to receive CPAP therapy
* informed consent

Exclusion Criteria:

* unstable angina or recent myocardial infarction (MI) (<4 weeks prior)
* severe valvular dysfunction
* requirement for revascularization
* a permanent pacemaker
* atrial fibrillation
* significant ventricular arrhythmia or sinus node dysfunction
* life expectancy less than 1 year due to other co-morbidity
* significant restrictive and obstructive lung disease
* concomitant treatment or use of: tricyclic antidepressants, cocaine or drugs which may alter catecholamine uptake; or hypnotic, benzodiazepine, selective serotonin reuptake inhibitors(SSRI), neuroleptic, narcotic or other medications which may alter sleep or sleep-disordered breathing
* central sleep apnea
* other primary sleep disorder (i.e. periodic limb movement with arousal >5 events/hr, narcolepsy, rapid eye movement (REM) behaviour disorder)
* requiring supplemental oxygen therapy at night
* debilitating daytime somnolence (indicating clear-cut indication for CPAP therapy)
* a previous cardiac transplant
* a large transmural scar defined on previous perfusion imaging(severe resting perfusion defect (<50% uptake) occupying >25% of the LV)148-150
* age < 18 years
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Measurements of oxidative metabolism (11C clearance rate constant 'k') and WMI | at 6-8 weeks
  The differences in the measurements of oxidative metabolism (11C clearance rate constant 'k') and WMI will be analyzed using t-tests for the treatment groups
C-11 Hydroxyephedrine (HED) retention | 6-8 weeks
  C-11 HED retention will be a measure myocardial SN pre-synaptic function in treatment groups

SECONDARY OUTCOMES:
Changes in other parameters including New York Heart Association (NYHA) class, HR, BP, LV volumes, stroke work-index, and QoL scores will also be analyzed. The subgroups of ischemic and non-ischemic etiology will be analyzed | at 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob S Beanlands, MD, FRCP C, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Hall AB, Ziadi MC, Leech JA, Chen SY, Burwash IG, Renaud J, deKemp RA, Haddad H, Mielniczuk LM, Yoshinaga K, Guo A, Chen L, Walter O, Garrard L, DaSilva JN, Floras JS, Beanlands RS. Effects of short-term continuous positive airway pressure on myocardial sympathetic nerve function and energetics in patients with heart failure and obstructive sleep apnea: a randomized study. Circulation. 2014 Sep 9;130(11):892-901. doi: 10.1161/CIRCULATIONAHA.113.005893. Epub 2014 Jul 3. PMID 24993098
- [Background] Johnson CB, Beanlands RS, Yoshinaga K, Haddad H, Leech J, de Kemp R, Burwash IG. Acute and chronic effects of continuous positive airway pressure therapy on left ventricular systolic and diastolic function in patients with obstructive sleep apnea and congestive heart failure. Can J Cardiol. 2008 Sep;24(9):697-704. doi: 10.1016/s0828-282x(08)70668-8. PMID 18787720
- [Background] Yoshinaga K, Burwash IG, Leech JA, Haddad H, Johnson CB, deKemp RA, Garrard L, Chen L, Williams K, DaSilva JN, Beanlands RS. The effects of continuous positive airway pressure on myocardial energetics in patients with heart failure and obstructive sleep apnea. J Am Coll Cardiol. 2007 Jan 30;49(4):450-8. doi: 10.1016/j.jacc.2006.08.059. PMID 17258090